CLINICAL TRIAL: NCT06451848
Title: A Single Center, Randomized, Double-blind, Single Dose Bioequivalence Trial of Genakumab in Chinese Healthy Male Adults
Brief Title: A Bioequivalence Study of Two Different Dosage Form of Genakumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GenSci048-104
Record Dates: First submitted 2024-05-28; First posted 2024-06-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-11

CONDITIONS: Gouty Arthritis (GA)
MeSH Terms: conditions — Arthritis, Gouty | interventions — Solutions; Injections; Powders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test preparation（T） (Experimental): Genakumab Solution for Injection (T, liquid formulation)
  Interventions: Drug: Genakumab Injection (T, Solution for injection); Drug: Genakumab for Injection (R, Powder for solution for injection)
- Reference preparation（R） (Experimental): Genakumab Powder for solution for Injection (R, lyophilized formulation)
  Interventions: Drug: Genakumab Injection (T, Solution for injection); Drug: Genakumab for Injection (R, Powder for solution for injection)

INTERVENTIONS:
Drug: Genakumab Injection (T, Solution for injection) — A single dose of subcutaneous injection of Genakumab（Solution for injection, liquid formulation）200 mg on Day 1
Drug: Genakumab for Injection (R, Powder for solution for injection) — A single dose of subcutaneous injection of Genakumab（Powder for solution for injection, lyophilized formulation) 200 mg on Day 1

SUMMARY:
The purpose of this study is to investigate whether Genakumab Injection is bioequivalent to Genakumab for Injection.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male aged ≥18 years old and≤45 years old;
* The Body mass index (BMI): 19-26 kg/m2 (inclusive), and body weight ≥50 kg;
* Subjects who voluntarily signed the informed consent form (ICF)；
* Subjects of childbearing potential had no plans for pregnancy or donating sperm/ova and agreed to use reliable contraception during the study and for 3 months after the last dose;

Exclusion Criteria:

* (During screening) Allergic to the investigational product, any of its components, or any biological agents, or had a history of multiple allergies (two or more) to drugs, foods, or environmental factors, or were prone to allergic symptoms such as rashes or urticaria;
* (During screening inquiry) Previously unable to tolerate intravenous puncture/indwelling needles for blood collection, or had a history of hemophobia or fear of needles;
* Abnormal vital signs (pulse < 50 bpm or > 100 bpm when awake, systolic blood pressure ≥ 140 mmHg or < 90 mmHg or diastolic blood pressure ≥ 90 mmHg or < 60 mmHg, forehead temperature > 37.3°C); ECG QTc-F interval ≥ 460 ms, or other clinically significant ECG abnormalities; abnormal findings in physical examination, laboratory tests, chest CT, and abdominal B-mode ultrasound;
* Subjects who have positive results of human immunodeficiency virus antibodies (HIV-Ab), or hepatitis B surface antigen (HBsAg), or hepatitis C virus antibodies (HCV-Ab), or syphilis specific antibodies (TPPA)；
* (During screening/admission inquiry) Had a clear history of neurological or psychiatric disorders (including epilepsy, dementia, depression, bipolar affective disorder, schizophrenia, etc.); history of prolonged QTc interval; immunodeficiency or immunosuppressive diseases, malignant tumors; clinically significant chronic diseases related to cardiovascular, liver, kidney, endocrine, respiratory, hematological (including coagulation), or digestive systems;
* Underwent major surgery (such as coronary artery bypass graft, liver or kidney resection, gynecological surgeries, etc.) within 6 months prior to the first dose; experienced acute neurological, digestive, respiratory, circulatory, endocrine, or hematological diseases within 3 months prior to screening that could affect the absorption, distribution, metabolism, excretion, and safety evaluation of the investigational product;
* History of drug abuse within 1 year prior to the first dose, or tested positive in a multi-drug urine test at admission；
* Smoked more than 5 cigarettes per day on average in the 3 months prior to screening or unable to cease use of any tobacco products (including nicotine products) during the study;
* Alcoholic or drank more than 14 units of alcohol per week in the 4 weeks prior to screening (1 unit equals 17.5 mL or 14g of pure alcohol. The alcohol content of different types of alcoholic beverages is indicated by volume percentage. One alcohol unit is approximately equivalent to 35 mL of 50% alcohol by volume [ABV] Baijiu or 350 mL of 5% ABV beer), unwilling to abstain from drinking alcohol or consuming any alcohol-containing products during the study, or tested positive for alcohol at admission;
* Received treatment with the investigational product or medical device in any clinical trial within 3 months prior to the first dose;
* Regularly used any prescription or over-the-counter (OTC) drugs, biologics, Chinese patent drugs, herbal supplements, vitamins, dietary supplements, or maintenance products within 2 weeks prior to the first dose, except for oral or implanted long-acting contraceptives;
* The investigator assessed that there were other factors making the subject unsuitable for participation in the study.etc.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 178 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (Area under the concentration-time curve (AUC), of Genakumab Injection with Genakumab for Injection | 0 hours -3360 hours post-administration
Pharmacokinetics (Peak Plasma Concentration (Cmax)）of Genakumab Injection with Genakumab for Injection | 0 hours -3360 hours post-administration
Pharmacokinetics (Peak time (Tmax) of Genakumab Injection with Genakumab for Injection | 0 hours -3360 hours post-administration
Pharmacokinetics (The elimination half-life (T1/2) of Genakumab Injection with Genakumab for Injection | 0 hours -3360 hours post-administration

SECONDARY OUTCOMES:
Safety and tolerability（Number of participants with treatment-related adverse events） | up to approximately 85 days

OTHER OUTCOMES:
Anti-drug antibody (Number of Participants with positive ADA) | 0 hours -3360 hours post-administration

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu Xinhua Hospital, Chengdu, Sichuan, China